CLINICAL TRIAL: NCT02759965
Title: Neuroinflammation and Cognitive Dysfunction After Orthopedic Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lars I Eriksson, Professor, Karolinska University Hospital
Other Study IDs: NEUPORT
Record Dates: First submitted 2014-11-10; First posted 2016-05-03 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Surgery; Acute Phase Reaction
MeSH Terms: conditions — Acute-Phase Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary hypothesis that orthopaedic surgery induces a neuroinflammatory response within 48 hours after elective hip or knee surgery and that there is an association between exaggerated CNS inflammatory response or impaired inflammatory resolution and postoperative cognitive dysfunction within one week and at three months postoperatively.

DETAILED DESCRIPTION:
Patients at 50-85 years of age undergoing orthopedic surgery will be investigated in the perioperative period to detect signs of neuroinflammation using serial CSF and blood sampling for 48 hours in combination with cognitive testing preoperatively, at 3-7 days and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Health Class 1-4
* Age 50-85 years
* Fluent in Swedish language
* Scheduled for primary hip replacement surgery due to arthrosis
* MMSE (minimental state test score >= 25.

Exclusion Criteria:

* Patient refusal to participate in the trial
* Current autoimmune disease, including arthritis
* Ongoing smoking, snuff or other nicotine compound treatment
* Significant neurologic or psychiatric disorder (such as Alzheimer's disease, Parkinson's disease, Multiple sclerosis, schizophrenia, depression, diagnosis of dementia or cognitive impairment as defined by a preoperative MMSE score ≤ 24
* History of stroke with neurological sequelae.
* Current severe cardiac (NYHA>IV) or renal (plasma creatinine> 0.250 mmol/l) Coagulopathy making spinal anesthesia and intrathecal catheter placement impossible
* Terminal phase of a chronic disease.
* Patient on chronic steroidal therapy
* Poorly controlled diabetes mellitus.
* Presumed uncooperativeness or legal incapacity.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 34 elective orthopedic patients undergoing hip or knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Neuroinflammation measured as IL-6 in CSF | Up to 48 hours postoperatively
  IL-6 in CSF

SECONDARY OUTCOMES:
Cognitive function | Before surgery, within 7 days after surgery and 3 month after surgery
  A cognitive test battery will be applied
Peripheral inflammatory response | Up to 48 hours
  Cytokines i peripheral blood
Neuroinflammation | Up to 48 hours
  CNS specific markers in blood
Neuroinflammation | Up to 48 hours postoperatively
  CNS specific markers in CSF
Neuroinflammation | Up to 48 hours postoperatively
  INflammatory Inflammatory markers in CSF

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Department of Anesthesiology, Surgical Services and Intensive Care Medicine, Karolinska University Hospital, Solna, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided